CLINICAL TRIAL: NCT01222143
Title: A Phase I/II Study Evaluating the Safety and Efficacy of Nilotinib Combined With Mitoxantrone, Etoposide, and High-Dose Cytarabine (NOVE-HiDAC) Induction Chemotherapy Followed by Consolidation Therapy for Poor-Risk Patients With C-kit Positive Acute Myeloid Leukemia (AML) up to Age 65
Brief Title: Safety and Efficacy Study of Nilotinib Combined With Mitoxantrone, Etoposide, and High-dose Cytarabine Induction Chemotherapy Followed by Consolidation for Patients With C-kit Positive Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107YCA03T
Record Dates: First submitted 2010-10-13; First posted 2010-10-18 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; NOVE-HiDAC; Nilotinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOVE-HiDAC and Nilotinib (Experimental): All patients will be receiving nilotinib combined with mitoxantrone, etoposide and high-dose cytarabine reinduction therapy. Patients achieving complete remission will receive consolidation therapy with nilotinib combined with high-dose cytarabine and mitoxantrone.
  Interventions: Drug: NOVE-HiDAC; Drug: Nilotinib

INTERVENTIONS:
Drug: NOVE-HiDAC — NOVE-HiDAC consists of mitoxantrone, etoposide, and modified high-dose cytarabine. During induction patients will receive mitoxantrone by IV on Days 6-10, etoposide by IV on Days 6-10 and cytarabine by IV on Days 11-12.
  During consolidation patients will be receiving mitoxantrone by IV on Days 1-10 and cytarabine by IV on Days 6, 8 and 10.
Drug: Nilotinib — The dose of nilotinib will be determined according to a dose escalation design. There will be three dose levels used in the study.
  During induction, nilotinib will be given orally on Days 1-12.
  During consolidation, nilotinib will be given orally on Days 1-10.

SUMMARY:
This is a phase I/II open-label study that is evaluating the toxicity and efficacy of nilotinib combined with mitoxantrone, etoposide, and high-dose cytarabine (NOVE-HiDAC) chemotherapy for patients with poor-risk acute myeloid leukemia (AML). There are two parts to the study. The first part (Phase I) will determine the maximum dose of nilotinib that can safely be given when combined with NOVE-HiDAC. This dose will then be used in combination with the NOVE-HiDAC regimen in the second part of the study (Phase II), which will evaluate the antileukemic activity of the treatment. The patients who achieve complete remission from the induction therapy (1 cycle) will then receive consolidation therapy combined with nilotinib (maximum of 2 cycles).

The patient population for this study will have AML and will fall into a poor risk category. This means they have persistent leukemia after induction therapy, they relapse within two years of achieving complete remission with induction therapy, or they have certain poor risk features at diagnosis. The AML cells will also be positive for c-kit (a stem cell factor receptor), which is involved in cancer cell growth. Nilotinib is a drug that blocks the effects of c-kit. Using this drug in combination with chemotherapy may improve ability of the chemotherapy drugs to kill leukemia cells. This may then increase the chances of the leukemia going into complete remission.

ELIGIBILITY:
Inclusion Criteria:

* AML as defined by WHO (World Health Organization) criteria, all subtypes except APL (acute promyelocytic leukemia).
* One of the following poor risk features:

  1. Persistent leukemia (at least 10% bone marrow blasts) after induction therapy, consisting of cytarabine 100-200 mg/m2 plus an anthracycline.
  2. Relapse within two years of achieving complete remission with such induction therapy. Any consolidation therapy is acceptable, including stem cell transplantation.
  3. No prior inductions, but antecedent myeloproliferative disorder or CMML (chronic myelomonocytic leukemia) (These patients are given NOVE-HiDAC as frontline therapy at Princess Margaret Hospital).
* Positivity for c-kit (CD117) in at least 30% of blasts as measured by flow cytometry. For relapsed patients, this will be assessed at the time of relapse. For primary induction failures the initial diagnostic sample may be used.
* Age 18-65.
* ECOG performance status < 3 (see Appendix I).
* Patients must have the following laboratory values within normal limits (WNL) at the local institution lab or corrected to WNL with supplements prior to first dose of study medication.

  1. Potassium (WNL)
  2. Magnesium (WNL)
* No chemotherapy within the previous four weeks, other than hydroxyurea to control counts. Hydroxyurea may be continued up to Day 4 of treatment with nilotinib. If hydroxyurea is used, it must be stopped at least 48 hours prior to starting chemotherapy.
* Able to give informed consent.

Exclusion Criteria:

* Active uncontrolled infection.
* Active CNS (central nervous system) leukemia
* Serum creatinine > 200 umol/L.
* Serum bilirubin > 1.5 x ULN, AST (aspartate aminotransferase) or ALT (alanine aminotransferase) > 2x ULN (upper limit of normal).
* Serum amylase and lipase > 1.5x ULN
* Left ventricular ejection fraction < 50%
* Impaired cardiac function including any of the following:

  1. Long QT syndrome or a known family history of long QT syndrome
  2. History or presence of clinically significant ventricular or atrial tachyarrhythmias
  3. Clinically significant resting bradycardia (< 50 beats per minute)
  4. Inability to monitor the QT interval by ECG
  5. QTc > 450 msec on baseline ECG (electrocardiogram). If QTc > 450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
  6. Myocardial infarction within 1 year of starting study drug
  7. Other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension)
* Patients currently receiving treatment with strong CYP3A4 inhibitors as listed in Section 5.8 and treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug
* History of acute or chronic pancreatic disease.
* Women who are pregnant, breast feeding, or of childbearing potential without a negative serum test at baseline. Male or female patients of childbearing potential unwilling to use contraceptive precautions throughout the trial and 3 months following discontinuation of study drug. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential must have a negative serum pregnancy test prior to the first dose of nilotinib.
* Known hypersensitivity to study drugs or other components.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of nilotinib when combined with the NOVE-HiDAC regimen (mitoxantrone, etoposide, and modified high-dose cytarabine). | 2 years
  To determine the maximum tolerated dose (MTD) of nilotinib combined with mitoxantrone, etoposide, and modified high-dose cytarabine (NOVE-HiDAC) induction chemotherapy followed by consolidation chemotherapy for patients with poor risk c-kit positive AML.
To evaluate the toxicity of the treatment regimen. | 2 years
To determine the complete response (CR) rate of this combination at the maximum tolerate dose (MTD) of nilotinib. | 2 years

SECONDARY OUTCOMES:
To determine the disease-free survival of this combination. | 2 years
To evaluate the pharmacodynamic effects of nilotinib on pERK and pAKT (phosphorylated ERK and AKT) in AML cells in vivo. | 2 years
To correlate clinical responses with the degree of pAKT and pERK inhibition achieved in vivo. | 2 years
To correlate the degree of pAKT and pERK inhibition with nilotinib pharmacokinetics. | 2 years
To correlate pAKT and pERK inhibition with c-kit mutations. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Brandwein, MD, FRCPC, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada